CLINICAL TRIAL: NCT04869839
Title: Oral Functions and Malocclusions: a Comprehensive Epidemiological Study on 358 Schoolchildren in France
Brief Title: Oral Functions and Malocclusions
Acronym: MALODYS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21Odonto01
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2021-04

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion | interventions — Diagnosis, Oral

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: oral examination — examination done by dentist

SUMMARY:
The aim of our research is to establish a link between malocclusions and oral dysfunctions. The clinical examination includes: caries screening (DMFT and dft scores), a quantification of dental plaque (Silness and Loë's plaque index) and orthodontic treatment need (Haute Autorité de Santé HAS). The functional examination includes improper mouth breathing, abnormal deglutition and incorrect position of tongue at rest.

ELIGIBILITY:
Inclusion Criteria:

* All the pupils benefit from the clinical examination

Exclusion Criteria:

* NONE

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Comprehensive study involving all six-grade schoolchildren in Cagnes sur mer, Alpes Maritimes, France
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Dental malocclusion - extraoral examination | 1 day
  Dental malocclusion as defined by the HAS:
  - An extraoral examination: sub-nasal profile, the sub-nasal angle and the labial-mental groove;
Dental malocclusion - intraoral examination | 1 day
  Dental malocclusion as defined by the HAS:
  - An intraoral examination: right and left molar dental class (Angle classification, overjet (abnormal when> 3mm)
Dental malocclusion - intraoral examination | 1 day
  Dental malocclusion as defined by the HAS:
  , number of patient with shifted midlines ,
Dental malocclusion - intraoral examination | 1 day
  Dental malocclusion as defined by the HAS:
  number of patient with an overbite (overbite> 2mm)
Dental malocclusion - intraoral examination | 1 day
  Dental malocclusion as defined by the HAS:
  number of patient with an open bite (overbite <0)

SECONDARY OUTCOMES:
Functional oral examination - ventilation | 1 day
  The functional pral examination includes improper mouth breathing: type of ventilation -1:
  Number of patient with adenoid facies
Functional oral examination - ventilation | 1 day
  The functional examination includes improper mouth breathing: type of ventilation - 2 Number of patient with a positive Glaze's test
Functional oral examination - ventilation | 1 day
  The functional examination includes improper mouth breathing: type of ventilation - 3 Number of patient with a positive Rosenthal's test
Functional oral examination - deglutition | 1 day
  The functional examination includes abnormal deglutition. Number of patient with an abnormal déglutition (clinical exam)
Functional oral examination - position of tongue | 1 day
  The functional examination includes i incorrect position of tongue at rest. number of patient with en incorrect position of the tongue (clinical exam)
Oral health | 1 day
  * Index of the severity of the caries disease (DMFT and dft);
  * Silness and Loë's plaque index (0: absence of plaque, 1: plaque not visible to the naked eye but detachable with the probe; 2: plaque visible to the naked eye; 3: abundant plaque visible to the naked eye in the sulcus and on the marginal gingiva)

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No